CLINICAL TRIAL: NCT01891825
Title: Persistent Atrial Fibrillation Ablation Trial
Acronym: PAAT
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Internal protocol review
Sponsor: Neil Sulke (Other)
Responsible Party: Sponsor-Investigator, Neil Sulke, Principal Investigator, Eastbourne General Hospital
Organization: Eastbourne General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PAAT
Record Dates: First submitted 2013-06-29; First posted 2013-07-03 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2014-06

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; Persistent atrial fibrillation; Atrial fibrillation ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pecutaneous AF ablation (Active Comparator): Percutaneous catheter ablation of atrial fibrillation
  Interventions: Procedure: Percutaneous AF ablation
- Surgical AF ablation (Active Comparator): Minimally invasive thoracoscopic surgical ablation of atrial fibrillation
  Interventions: Procedure: Surgical AF ablation

INTERVENTIONS:
Procedure: Surgical AF ablation — Minimally invasive thoracoscopic surgical ablation of atrial fibrillation
  Arms: Surgical AF ablation
Procedure: Percutaneous AF ablation — Percutaneous catheter ablation of atrial fibrillation
  Arms: Pecutaneous AF ablation

SUMMARY:
Persistent atrial fibrillation (AF) is a common and distressing condition, that can cause significant symptoms. AF ablation is a recognised technique to treat persistent AF, but can be technically difficult. This study compares percutaneous ablation to thoracoscopic surgical AF ablation.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic persistent or long-standing AF suitable for AF ablation.
* Age over 18 years old.
* Informed consent to participate in this study.

Exclusion Criteria:

* Pre-existing ILRs or permanent pacemakers that do not allow for continuous monitoring for AF occurrence, or are not MRI-safe.
* Unable to undergo general anaesthesia for AF ablation.
* Previous cardiac surgery, such as coronary artery bypass grafting or valvular surgery.
* Scheduled for elective cardiac surgery, such as coronary artery bypass grafting or valvular surgery.
* Previous thoracic surgery.
* Participation in a conflicting study.
* Potential participants who are mentally incapacitated and cannot consent or comply with follow-up
* Pregnancy
* Other cardiac rhythm disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-09; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Recurrence of persistent AF by 12 months after ablation | 12 months
  Mean time to recurrence of persistent AF after ablation

SECONDARY OUTCOMES:
Change in AF burden after AF ablation | 12 months
  Detected by ILR
Time to first episode of symptomatic AF after ablation | 12 months
  Time to first episode of symptomatic AF after ablation
Time to first episode of any AF after ablation | 12 months
  As detected by ILR
Total number of AF episodes after AF ablation | 12 months
  As detected by ILR, outside blanking period
Total number of AF episodes lasting greater than 6 minutes after AF ablation | 12 months
  As detected by ILR, outside blanking period
New MRI-detected subclinical cerebral embolic events | 3 months

OTHER OUTCOMES:
Quality of life changes after AF ablation | 12 months
Change in exercise capacity assessed by cardiopulmonary exercise testing (CPET) after AF ablation | 12 months
Change in echocardiographic left atrial dimensions and function after AF ablation | 12 months
Change in cognitive function as assessed by the Mini Mental State Examination (MMSE) and Montreal Cognitive Assessment (MoCA) instruments | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Neil Sulke, DM, Principal Investigator — Eastbourne General Hospital
Locations (2):
- United Kingdom (2):
  - Eastbourne General Hospital, Eastbourne, E Sussex
  - Royal Sussex County Hospital, Brighton, East Sussex